CLINICAL TRIAL: NCT03864471
Title: Evaluation of a Care Delivery Model for the High-need Community Older Adults
Brief Title: High-need Community Older Adults Care Delivery Model
Acronym: HCOACDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuei-Min Chen, Ph.D., RN., Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KMUHIRB-F(I)-20170070
Record Dates: First submitted 2019-03-02; First posted 2019-03-06 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: High-need Older Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCOACDM (Experimental): The intervention, the HCOACDM, involves case screening, comprehensive assessment, and care coordination, and will be given over a 6-month period.
  Interventions: Other: HCOACDM
- Routine care (Active Comparator): The routine care services include home visits, telephone checkups, meals on the wheel, and health promotion activities.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: HCOACDM — The intervention, the HCOACDM, involves case screening, comprehensive assessment, and care coordination, and will be given over a 6-month period.
  Arms: HCOACDM
Other: Routine care — The routine care services include home visits, telephone checkups, meals on the wheel, and health promotion activities.
  Arms: Routine care

SUMMARY:
This study is proposed to: (1) establish a "High-need Community Older Adults Care Delivery Model" (HCOACDM) as a guide to handle complex needs of the high-need community older adults by the care managers at community care centers; and (2) evaluate the effectiveness of applying the HCOACDM to improve the functional ability, quality of life (QOL), depressive symptoms, healthcare and social service utilizations, and care delivery satisfaction of the high-need community older adults.

DETAILED DESCRIPTION:
A cluster randomized controlled trial with repeated measures design will be conducted to test the effectiveness of six-month HCOACDM on the functional ability, QOL, depressive symptoms, healthcare and social service utilizations, and care delivery satisfaction of the high-need community older adults. The high-need community older adults, screened based on the "High-need Community Older Adults Screening Scale" (HCOASS), will be cluster randomized based on the community care centers, to the intervention group (4 centers) or comparison group (4 centers). Intervention group will receive six-month HCOACDM care and comparison group will receive original routine care provided by the care managers at community care centers. One pre-test and two post-tests, three months apart, of outcome measurements will be conducted on all participants. Moreover, individual semi-structured interviews will be carried out to explore opinions and suggestions toward the HCOACDM of the care managers in intervention group. It is expected that the developed HCOACDM will be useful to provide the long-term care for community older adults and enhance the quality of diverse and complex care delivery system.

ELIGIBILITY:
Inclusion Criteria:

* lived in the community at least three months
* over 65 years old
* fluently communicated in Mandarin or Taiwanese
* screened by the High-need Community Older Adults Screening Scale (HCOASS) as high-need older adults

Exclusion Criteria:

* diagnosed as dementia

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 165 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Functional Ability measured by the Barthel Index (BI) | 6 months
  A 10-item scale that includes feeding, transfers, grooming, toilet use, bathing, mobility, stairs, dressing, and control of bladder and bowel. Score ranges from 0 to 100; the higher the score, the higher the level of self-care independence of an individual: 0-20 = complete dependence, 21-60 = severe dependence, 61-90 = moderate dependence, 91-99 = mild dependence, and 100 = total independence.
Quality of Life measured by the World Health Organization quality of life (WHOQOL-BREF) | 6 months
  A 28-item scale with four dimensions: physical health, psychological health, social relations, and environment. The responses use a 5-point Likert scale; the higher the score, the better the QOL of an individual.
Depressive Symptoms measured by the Hamilton Depression Rating Scale (HDRS) | 6 months
  A 17-item scale uses to assess a client's emotional and physical-psychological status during the past week through a self-report and observations. The total score ranges from 0 to 52: a score > 18 = severe depression, 14-17 = moderate depression, 11-13 = mild depression, 8-10 = borderline depression, and < 7 as normal.

SECONDARY OUTCOMES:
Healthcare and Social Service Utilizations measured by the Resource Usage of the High-concerned Community Older Adults | 6 months
  Based on the long-term care services that are provided in Taiwan, 21 resources are itemized in 3 categories: 1) care for the client (8 services), 2) social welfare (10 services), and 3) care for the caregiver (3 services). The researcher will mark the services that have been used by the participants.
Satisfaction with Care Delivery measured by the Satisfaction Questionnaire of Service Users to Care Managers | 6 months
  There are three dimensions in the questionnaire (Chiou, 2011), but only the dimensions of professional abilities (5 items) and interpersonal interactions and attitudes (5 items) are adopted in this study. A 5-point Likert scale is used; the higher the score, the more satisfaction a client has with the service provider.

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Min Chen, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Community Care Centers, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No